CLINICAL TRIAL: NCT03531164
Title: Effect of Kayak Ergometer Training in Trunk Control, Independence and Cardiovascular Health in Individuals With Spinal Cord Injury
Brief Title: Kayak Ergometer Training in Individuals With Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Jimena Quinzaños, MD, MSc, Instituto Nacional de Rehabilitacion
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 74/15
Record Dates: First submitted 2018-03-05; First posted 2018-05-21 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injuries; kayak; trunk control
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kayak ergometer group (Experimental): Intervention: Training in kayak ergometer: 3 minutes of warming (pre-charge) , 3-5 intervals of training with moderate to high intensity and pauses of 2-4 minutes (charge) and 2 minutes of cooling down (post-charge) to complete 30 minutes.
  Interventions: Other: kAYAK ERGOMETER GROUP
- Control group (Active Comparator): Intervention: 30 minutes of proprioceptive neurofacilitation focused on trunk control
  Interventions: Other: CONTROL GROUP

INTERVENTIONS:
Other: kAYAK ERGOMETER GROUP — Kayak ergometer training for 30 min 5 times a week for 6 weeks. The training includes a warming (pre charge) during 3 minutes, a training (charge) characterised by 3-5 intervals with medium to high intensity during 2-4 minutes and pauses of 1-2 minutes between active phases and 2 minutes of cooling down (post charge) to complete 30 minutes of training.
  Arms: Kayak ergometer group
Other: CONTROL GROUP — Proprioceptive neurofacilitation exercises focused in trunk control during 30 minutes 5 times a week for 6 weeks.
  Arms: Control group

SUMMARY:
One of the main objectives in spinal cord injury rehabilitation programs is the improvement of trunk control in order to achieve independence, to prevent complications and, in specific cases to walk.

Research question: What is the effect of kayak ergometer training in trunk control, cardiovascular condition and independence in individuals with a spinal cord injury? Purpose: To determine the effect of kayak ergometer training in trunk control, cardiovascular condition and independence in individuals with a spinal cord injury.

Methods: Randomized clinical trial, blinded to evaluator and to the person that will analyze data.

Population: Spinal cord injured individuals treated at the National Institute of Rehabilitation, with a spinal cord injury of any ethiology, with a neurologic level of C8 and below, with time since injury from three months to one year.

Proceeding: The subjects will be randomly assigned to : a control group with neuro propioceptive facilitation exercises focused in trunk control or an experimental group with kayak ergometer training. Both groups will recieve 5 sessions a week during 6 weeks.

DETAILED DESCRIPTION:
Spinal Cord Injury (SCI) is an alteration of the spinal cord that modifies not only muscular strength and sensitivity, but that also generates a change in all of the systems of the organism. At the worldwide level, an incidence is calculated of between 13.1 and 52.2 per one million inhabitants.

Damage to the ascending and descending tracts of the spinal cord consequently gives rise to an alteration in the postural control system. It is known that effective postural control is of utmost importance forstanding and walking, as well as for providing support for voluntary movements. Alterations in posture depend on the grade and level of the injury; thus, persons with complete, thoracic, or cervical lesions have poor trunk control. Due to the latter, they are limited in many of the movements necessary for carrying out daily life activities (DALYS) Therefore, part of the objectives of rehabilitation in individuals with an SCI comprises improvement in trunk control.

On the other hand, patients with SCI tend to engage in a sedentary lifestyle that, added to the alterations in the autonomic nervous system proper to the lesion, exposes individuals with a SCI to a greater risk of developing chronic-degenerative conditions, such as metabolic syndrome and cardiovascular diseases, which are, at present, the main cause of death in these persons.

Thus, after the immediate rehabilitation, it is necessary to maintain and improve the functional capacity obtained during this process. Therefore, it is important to find training activities to challenge stabilization of the upper part of the body and sitting equilibrium without giving rise to symptoms caused by overuse.

Kayak training appears to comply with these criteria, in that it implicates the greater part of the upper musculature, presents high metabolic demands, and imposes strict requirements for the balance control system, due to continuous compensation of the disturbances of the upper part of the body caused by movement on the apparatus. It was previously demonstrated that open-sea training in kayaks could be implemented in a group of individuals in paraplegic condition and that this is accompanied by improvements in strength and equilibrium in sedestatIon.

Due to the difficulty in controlling and adjusting the time and challenge level of the equilibrium experienced by participants at sub-acute stages, it is necessary to utilize a kayak ergometer, in such a way that the demand for equilibrium can be adjusted individually and for this to increase progressively as the treatment advances. In this respect, Bjerkefors and Thorstensson demonstrated that kayak ergometer training in a group of persons with SCI is accompanied by improvement in shoulder muscular strength and in various functional wheelchair tests that demand trunk stabilization and balance control.

These studies achieved demonstrating the positive effect of kayak training in patients with SCI; however, in these studies, small populations were included (10 and 12 individuals), with chronic-stage lesions, and the effects on trunk control were not evaluated by means of a validated scale in this population, nor were the training's effects on cardiovascular function and functional independence.

To date, the effect of kayak ergometer training has not, to our knowledge, been studied in individuals with SCI in terms of trunk control with tools validated for persons with SCI, regarding the cardiovascular condition, functional independence, and quality of life, thus engendering the need to conduct this present study.

HYPOTHESIS

Kayak ergometer training will improve functional independence, trunk control, and cardiovascular condition in individuals with SCI.

The effect of training with the kayak ergometer on functional independence, trunk control, and the cardiovascular condition in individuals with SCI will be greater than that of conventional trunk-control training.

GENERAL OBJECTIVE

To determine the effect of kayak ergometer training in patients with SCI in functionality, trunk control, cardiovascular condition, and quality of life.

SPECIFIC OBJECTIVES

* Establish the validity, reliability, error, and sensitivity of the measurement instrumented of trunk control in subjects with SCI.
* Evaluate the existence of floor/ceiling effects in the instrumented assessment of trunk control.
* Develop computerized tools for evaluation of trunk control that are easily applicable in daily clinical practice, with low-cost, practical, and simple technology for improving the exactness and reliability of the observational analysis, for rehabilitation centers that are not equipped with a movement-analysis laboratory, with sufficient information for evaluating the trunk control of the individual with SCI.
* Proposal of a pilot program of trunk control rehabilitation in persons with SCI.
* Broadcast preliminary results at a national scientific meeting.
* Form human resources with knowledge of neurological rehabilitation, movement analysis, and biomedical engineering.
* Foster multidisciplinary cooperation.

MATERIALS AND METHODS

Study type. Randomized controlled clinical trial blinded to the evaluator and to the person performing the data analysis.

Description of the work universe. Patients of out-patient consultations and hospitalization of the SCI Service of the National Institute of Rehabilitation), with a diagnosis of SCI of any etiology, with a neurological level of under C8, with a SCI of 3 months of evolution.

Definition of the control group Group A. Control group, management with conventional therapy for improvement of trunk control (proprioceptive neurofacilitation exercises focused on trunk control21) of 20 minutes five times weekly during 6 weeks.

Sample size We utilized the Epidat ver. 4 statistical software program to calculate sample size. For 80% study power and an alpha error probability of less than 0.05, and considering the work of Grigorenko and collaborators18 we found a frontal displacement speed difference of the Center of Pressure (CoP) of 0.1m/s with a Standard Deviation (SD) of 0.05 m/s between the experimental and the control group. Therefore, seven patients per group were required. Considering a possible loss of 20%, we will recruit nine patients per group.

Description of the study variables, units of measure, and measuring scales

Clinical and demographic variables

* SCI severity: According to American Spinal Injury Association, with International standards for neurological classification of spinal cord injury modifications: complete, B: incomplete, preservation of only the sensitive function, C: incomplete, voluntary anal contraction or more than half of key muscles in <3, D: incomplete, more than half of the key muscles in >3, E: total recuperation A, B, C, D, E
* Neurological level: More caudal segment of the SC with normal function
* Time of evolution of the SCI:Time in days elapsed from when the SCI was produced until time of application of the questionnaire
* Age:Years elapsed from date of birth to time of questionnaire application

Proposed statistical analysis

The investigators will utilize the Statistical Package for the Social Sciences ver. 17 statistical software program. The investigators will perform descriptive statistics with central-tendency measurements for quantitative variables and with proportions for qualitative variables. To determine differences between groups, analysis of covariance will be carried out. Results that are statistically significant with a p of <0.05 will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of spinal cord injury with any American Spinal Injury Association Impairment Scale (AIS) classification
* Neurologic level below C8
* Time since injury form 3 to 12 months
* Any aetiology

Exclusion Criteria:

* Another neurologic diagnosis
* Sense organ alteration
* Orthopaedic problem that interferes with training
* Alteration in superior mental function
* Cardiovascular or metabolic disease that interferes with trainig

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Trunk control | 6 weeks
  Score between 0-24, cut-off point 13. Higher values represent better results. The clinical trunk control test for individuals with spinal cord injury will be used

SECONDARY OUTCOMES:
Spinal Cord Injury Independence Measure III | Before training
  Validated specific independence measure for spinal cord injury. The main domains will be contemplated as secondary outcomes (Catz A, Spinal Cord 2007). Score ranges between 0 and 100. Higher values represent better results.
Spinal Cord Injury Independence Measure III | 6 weeks
  Validated specific independence measure for spinal cord injury. The main domains will be contemplated as secondary outcomes (Catz A, Spinal Cord 2007). Score ranges between 0 and 100. Higher values represent better results.
Cardiac frequency | Before training
  Registered with a polar
Cardiac frequency | 6 weeks
  Registered with a polar
Arterial tension | Before training
  Registered with a sphygmomanometer
Arterial tension | 6 weeks
  Registered with a sphygmomanometer
Satisfaction with life | Before training
  Life satisfaction questionnaire-9 is a validated questionnaire to assess life satisfaction in people with a spinal cord injury. It is composed of 9 questions that are rated by the patient between 1 (very dissatisfying) to 6 (very satisfying) and that explore perception in life as a hole, vocational, financial and leisure situations, contact with friends and acquaintances, sexual life and family life, partnership relation, physical and psychological health. Score ranges between 9 and 54. Higher values represent better results.
Satisfaction with life | 6 weeks
  Life satisfaction questionnaire-9 is a validated questionnaire to assess life satisfaction in people with a spinal cord injury. It is composed of 9 questions that are rated by the patient between 1 (very dissatisfying) to 6 (very satisfying) and that explore perception in life as a hole, vocational, financial and leisure situations, contact with friends and acquaintances, sexual life and family life, partnership relation, physical and psychological health. Score ranges between 9 and 54. Higher values represent better results.
Metabolic Equivalent of Task | Before training
  Exercise tolerance test
Metabolic Equivalent of Task | 6 weeks
  Exercise tolerance test
Oxygen consumption | Before training
  Exercise tolerance test
Oxygen consumption | 6 weeks
  Exercise tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: JImena Quinzaños, MD, MSc, Principal Investigator — Instituto Nacional de Rehabilitacion
Locations (1):
- Instituto Nacional de Rehabilitacion, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data base whithout identificatiopns
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After january 2022 for 5 years
Access Criteria: Ask the authors directly by mail